CLINICAL TRIAL: NCT00441428
Title: Safety And Efficacy Of Solifenacin In Men With Overactive Bladder (OAB) And Detrusor Underactivity
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Other Study IDs: UDASOL-1520
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Overactive Bladder; Detrusor Underactivity
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder, Underactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: solifenacin

SUMMARY:
Detrusor underactivity (DUA) in men is responsible for LUTS in a significant minority, the symptoms being indistinguishable from those seen in BOO. The International Continence Society (ICS) defines DUA as 'a detrusor contraction of inadequate magnitude and/or duration to effect complete bladder emptying in the absence of urethral obstruction. Whilst a reduced maximum urinary flow rate (Qmax) is indicative of voiding dysfunction, flow studies cannot distinguish between DUA and BOO, which are the two principal causes of low flow rates. DUA is diagnosed from a pressure-flow study (PFS)and is characterized by a low-pressure, poorly sustained, or wave-like detrusor contraction with an associated poor flow rate.

Overactive bladder (OAB) is the most common term currently used in clinical medicine to describe a complex of lower urinary tract symptoms (LUTS) with or without incontinence but most commonly consisting of urgency, frequency, nocturia, troublesome or incomplete emptying,and, occasionally, pain. With the exception of pain and incontinence, these symptoms are often found together; thus, the term LUTS has come to replace previous terms, such as urgency-frequency syndrome,urethral syndrome, and prostatism.

Drug treatment is frequently used as the initial management approach for LUTS in older men.Among men who desire treatment, general practice prescribing data have shown that antimuscarinics are not often given to elderly men. There is theoretical concern that the inhibitory effect of antimuscarinics on detrusor contraction could aggravate voiding difficulties or cause urinary retention in patients with BOO. There are virtually no data evaluating the safety and efficacy of solifenacin treatment in men with DUA and OAB.

ELIGIBILITY:
Inclusion Criteria:

* Men aged > 40 years were eligible if by 7-day bladder diary they had urinary frequency (8 or more micturitions per 24 hours) and urgency, with or without urgency incontinence (1 or more episodes per 24 hours) together with coexistence low detrusor contractility.

Exclusion Criteria:

* Urinary tract infection,
* Bladder stone, urogenital tumors,
* Prostate surgery,
* Use of indwelling catheter or self-catheterization program,
* Medications that could affect the lower urinary tract function,
* History of neurological disease,
* Acute urinary retention or any condition for which antimuscarinic was contraindicated.
* Antimuscarinic, antispasmodic, or electrostimulation within 1 month;
* Any investigational drug within 2 months; or
* A 5a-reductase inhibitor within 3 months of screening.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-02; Primary Completion 2007-01

PRIMARY OUTCOMES:
We estimated the safety of solifenacin treatment by measuring the changes to day 120 of voiding function. The following variables were assessed: BVE, BCI, BOOI, Qmax obtained during UDS, PVR

SECONDARY OUTCOMES:
We estimated the efficacy of solifenacin treatment. For this purpose, the primary efficacy measure was change in the number of urge incontinence episodes per week. Secondary efficacy measures included patient perception of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ronchi, M.D, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Abruzzo, Italy